CLINICAL TRIAL: NCT04116606
Title: A Randomised, Placebo-controlled, Double-blind Trial of the Antidepressant Efficacy of a Novel CNS-penetrant P2X7 Receptor Antagonist, JNJ-54175446, in People With Major Depressive Disorder, an Incomplete Response to Monoaminergic Antidepressant Drugs, and a Biomarker Profile Predictive of Active P2X7 Signalling
Brief Title: Antidepressant Trial With P2X7 Antagonist JNJ-54175446
Acronym: ATP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CCTU-Core (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, CCTU-Core, Chief Investigator, Cambridgeshire and Peterborough NHS Foundation Trust
Organization: Cambridgeshire and Peterborough NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCTU0251; 2018-001884-21 (EudraCT Number)
Record Dates: First submitted 2019-09-19; First posted 2019-10-04 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Depressive Disorder, Major; Inflammation
Keywords: P2X7; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active JNJ-54175446 (Active Comparator): JNJ-54175446 is an unlicensed drug currently being developed by Janssen Pharmaceuticals. The drug is presented in oral capsules, each capsule containing 50 mg of JNJ-54175446. Participants will be asked to self-administer one capsule daily for 8 weeks.
  Interventions: Drug: Active JNJ-54175446
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active JNJ-54175446 — JNJ-54175446 is a novel, potent, selective, and brain-penetrant antagonist of the adenosine triphosphate (ATP)-gated P2X7 channel.
  Arms: Active JNJ-54175446
Drug: Placebo — Matching placebo containing the same excipients
  Arms: Matching placebo

SUMMARY:
Depression is one of the most important causes of disability in the world today, with major personal, social and economic costs. Although some moderately effective drug treatments are already available, about a third of patients with major depressive disorder (MDD) remain depressed despite current treatment.

There is growing evidence that inflammation - the response of the body's immune system to physical and social stresses - can cause depressive symptoms in some patients. It is therefore predicted that anti-inflammatory drugs could have anti-depressant effects and the research team aims to test this using a new drug, JNJ-54175446, which blocks the activity of a receptor called P2X7. P2X7 is present on many immune cells and plays a key role in the release of inflammatory molecules during stress, which may be linked to stress-related depression.

The research team will recruit approximately up to 142 participants with MDD to this clinical trial. Patients will have moderate-severe depressive symptoms despite ongoing treatment with a conventional anti-depressant drug, and they will have blood test results at screening that indicate they are likely to have active P2X7 signalling in the brain. Eligible participants will be randomly allocated to receive either 50mg/day JNJ-54175446 or placebo for 8 weeks. Participants will be assessed at weeks 2, 5 and 8 using a standard clinical depression scale and the scores compared between those treated with placebo and those treated with JNJ-54175446. To understand more about the effects of JNJ-54175446 on the immune system and the brain, patients will also complete additional blood tests, questionnaires and magnetic resonance imaging (MRI) brain scans at different visits throughout the trial. The trial will be carried out across 5 centres in the UK.

DETAILED DESCRIPTION:
This trial will be a multi-centre, phase II, randomised, double blinded, placebo-controlled, parallel group trial.

The research team estimates that the majority of the participants will be recruited through the trial website, posters and research databases. In order to better assess the suitability of the interested participants, interested participants are required to answer pre-screening questions.

Only those who might be suitable to take part will be invited to a screening visit to continue with the rest of the trial screening procedures. The trial will consist of 3 phases - a screening phase, treatment phase of 8 weeks and follow up phase. This includes a total of 6 clinic visits and will be spread over about 15 weeks. Each clinic visit will last between 1.5 hours to 5 hours. Participants will have to be fasted overnight (10 hrs) prior to baseline visit 1 and visit 4 for biomarker blood samples. At these visits, breakfast will be provided after sample collection.

The list below outlines the study schedule and key assessments applicable to a participant who passes the pre-screening questions:

Screening phase clinic visit Participants who are interested in taking part will be invited to attend a screening visit in the clinic which lasts about 4 hours. At this visit the trial team will discuss the trial further and answer any queries the participants may have. If the participants agree, they will then provide informed consent prior to any screening tests and procedures being undertaken. An alcohol breath test and urine drug screen will be carried out. Urine samples will be taken for urinalysis.

Blood samples will be taken for safety assessments including full blood count, clinical chemistry tests, thyroid function tests, pregnancy and Follicle-stimulating hormone test (if applicable). Biomarker blood samples will also be taken for genetic analysis of P2X7 receptor and analysis of C-reactive protein (CRP) for eligibility check, and for other biomarker assays including genetic analysis. Other screening assessments include a review of the participant's medical and medication history, review of their depressive disorder and self-reported stress, and a physical examination. Vital signs will be measured and participants will have an electrocardiogram (ECG) performed. Participants will also be introduced to the other trial activities that will have to be carried out in their homes. This includes collection of saliva samples, the use of activity monitoring device and completion of daily sleep diary.

Screening phone call Once results from the genetic analysis of the P2X7 receptor and CRP levels are available (about 1 to 2 weeks after the screening visit), the results will be returned to the site team who will then inform the participant by phone whether they are eligible. If eligible, a baseline clinic visit will be arranged.

During this call, eligible participants will be reminded that saliva sample collection packs will be sent in the post, to collect saliva samples at specific time points and return them to the research team. Participants will also be sent an activity monitoring watch and sleep diary; participants should start wearing the watch everyday for at least 7 days prior to baseline visit and record their sleep.

Baseline/Treatment phase Visit 1 Participants will be asked to fast a minimum of 10 hours and attend a baseline site visit (Day 1) which would last approximately 5 hours.

At this visit, the participant's diagnosis of major depressive episode will be re-checked to ensure they are still eligible. Fasting blood samples will be taken for full blood count, clinical chemistry, biomarkers and baseline drug concentration analysis. After breakfast is given, an alcohol breath test and urine drug screen will be carried out. Urine samples will be taken for urinalysis and pregnancy test (if applicable). An ECG will be performed and vital signs will be assessed. Participants who continue to meet eligibility will be randomised in 1:1 ratio to receive JNJ-54175446 or placebo.

Participants will be asked about any adverse events and concomitant therapies. Various clinical and participant reported questionnaires will be completed to assess stress, depression symptoms and suicidal risk. Participants will be asked to complete a range of online cognition tests, during which heart rate variability measurements will be carried out. Participants will also have a baseline MRI scan which includes completion of a cognitive task during the scan. At the end of the visit, participants will receive 1 bottle of allocated trial drug and will be instructed to take 1 capsule every day within 30 minutes after breakfast. A medication diary will be provided to aid participants in recording their daily administration. Data from the activity watch will be downloaded and a new copy of daily sleep diary will be provided.

Visit 2 and Visit 3 Participants will be required to attend a visit to the site at Day 14 ± 2 (Visit 2) and at Day 32 ± 3 (Visit 3), each visit will last approximately 3 ½ hours. Participants do not need to be fasted for these visits. On these days, participants should not take their trial drug at home, they will be asked to take the drug at clinic after their blood and urine collection. At this visit, blood samples will be taken for full blood count, clinical chemistry analysis, CRP and drug concentration analysis. A urine drug screen will be carried out. Urine samples will be taken for urinalysis and pregnancy test (if applicable). Participants will then be asked to take their drug. An ECG will be performed and vital signs will be assessed. Participants will be asked about any adverse events and concomitant therapies. Various clinical questionnaires will be carried out to assess stress, depression and suicidal risk. Participants will be asked to complete a range of online cognition tests. Participant's trial drug compliance will be reviewed through review of the medication diary (visits 2 and 3) and physical counting of returned capsules (visit 3). Data will be downloaded from the activity monitoring device at each of these visits and a new daily sleep diary will be provided. At visit 3, participants will receive the 2nd bottle of allocated trial drug.

Telephone checks In order to maintain regular contact with the participants, the research team will contact the participants by telephone 8 to 12 days after visit 2 (phone check #1) and 8 to 12 days after visit 3 (phone check #2). Participants will be asked if they have had any adverse events, any changes to concomitant therapies and if they had been able to take the trial drug according to trial instructions.

At phone check #2, participants will also be instructed to collect saliva samples within 7 days before the next visit. The saliva collection packs will be posted to the participants.

Visit 4 Participants will attend a clinic visit on Day 56 ± 3 (Visit 4) lasting approximately 5 hours. Participants need to come to the site in fasted condition (minimum of 10 hours) and should not take their trial rug at home, they will be asked to take the drug at clinic after blood and urine collection and breakfast. This will be the final dose for the participants. At this visit, fasting blood samples will be taken for full blood count, clinical chemistry analysis, CRP and biomarkers and drug concentration analysis. A urine drug screen will be carried out. Urine samples will be taken for urinalysis and pregnancy test (if applicable). Participant will then be asked to take their drug. An ECG will be performed and vital signs will be assessed. Targeted physical examination will be carried out. Participants will be asked about any adverse events and concomitant therapies. Various clinical and participant reported questionnaires will be completed to assess stress, depression symptoms and suicidal risk. Participants will be asked to complete a range of online cognition tests, during which heart rate variability measurements will be carried out. The anti-depressant response will be assessed using a clinical scale (MADRS). Participants will also have a post-treatment MRI scan which includes completion of a cognitive task during the scan. Data will be downloaded from the activity monitoring device and the device collected from the participants. All unused drug will be collected from the participants.

Follow up visit (Visit 5) A follow-up visit will be scheduled between 7 and 14 days after last dose of administration (visit 4) and will last approximately 1 hour. Blood samples will be taken for full blood count, clinical chemistry and CRP analysis. Urine samples will be taken for urinalysis and pregnancy test (if applicable). An ECG will be performed and vital signs will be assessed. Participants will be asked about any adverse events and concomitant therapies. Targeted physical examination and medical review of symptoms and systems will be carried out and body weight measured. Participants will be asked to complete a depression questionnaire.

Home-based trial assessments Participants will be requested to wear the activity monitoring device from 7 days prior to visit 1 (Day -7) up until visit 4, and complete a daily sleep diary. This activity monitoring device will record the participant's activity and sleep patterns.

Participants have to self-administer 1 capsule of trial drug daily, preferably in the morning and within 30 min after breakfast. The date and time of administration should be recorded in the medication diary.

Participants will have to provide 2 sets of 6 saliva samples each during the trial.

Data analysis The primary endpoint is the change between baseline score and score at final dose on visit 4 (week 8) assessed by the MADRS scale. 142 participants will be enrolled. All data will be analysed and summarised in a clinical trial report.

ELIGIBILITY:
The key eligibility criteria are listed below, to obtain the full list please contact the trial team.

Inclusion Criteria:

1. Provided written informed consent
2. Between the age of 18 to 60 years inclusive
3. Meets the Diagnostic and statistical manual - 5 (DSM-5) diagnostic criteria for MDD without psychotic features (past or present), as confirmed by the M.I.N.I v7.0.
4. Has PHQ-9 score of ≥10.
5. BMI between 18.0 and 36.0 kg/m2 inclusive.
6. Currently being treated with one antidepressant monoaminergic drug (e.g. SSRI, SNRI, TCA) at an adequate dose, and for at least 6 weeks.
7. Must be medically stable based on clinical laboratory tests, medical history, vital signs, and 12-lead ECG performed.
8. Agree to practice highly effective method of birth control as stated in the protocol.
9. A woman of childbearing potential must have a negative serum pregnancy test at screening.
10. Agree not to donate eggs or sperm from start of dosing and for at least 3 months after receiving the last dose of study drug.

Exclusion Criteria:

1. Has a primary DSM-5 diagnosis of posttraumatic stress disorder.
2. Has failed to respond to more than 3 antidepressant treatments despite an adequate dose and duration, in the last 24 months.
3. Presence of two copies of the loss-of-function C allele at rs3751143, and/or has one copy of the loss-of-function A allele at rs1653624 in the P2RX7 gene.
4. Has a current or recent history of clinically significant suicidality.
5. Has a history of moderate or severe substance or alcohol use disorder according to DSM-5 criteria, except nicotine or caffeine, within 12 months before screening.
6. Has positive test result(s) for alcohol or drugs of abuse (including methadone, opiates, cocaine, cannabinoids, amphetamine/methamphetamine and ecstasy).
7. Has a current diagnosis of a psychotic disorder (e.g. schizophrenia, bipolar disorder), an eating disorder (e.g. anorexia, bulimia), or learning disability or a personality disorder that is considered by the investigator to interfere with the ability of the subject to adhere to the protocol (e.g. narcissistic personality, borderline personality disorder)
8. Has used:

   * Monoamine oxidase inhibitors (MAOIs) within 12 weeks before screening
   * Within 6 weeks prior to enrolment use of other antidepressant drugs not belonging to the allowed classes of SSRI, SNRI, or TCA.
9. Is currently treated with antipsychotic drugs (D2-antagonists; except for low-dose quetiapine), lithium, other mood stabilizers or opiates.
10. Unable to complete MRI scans.
11. Has current signs/symptoms of liver or renal insufficiency, diabetes mellitus (type I and II), hypothyroidism or hyperthyroidism without stable treatment, or other significant and uncontrolled medical conditions.
12. Is a woman who is pregnant or breast feeding.
13. Plans to conceive a child while enrolled in this study or within 3 months after the last dose of IMP.
14. Has a history of malignancy within 5 years before screening.
15. Has received an investigational drug/vaccines, used an invasive investigational medical device within 60 days before the planned first dose of IMP, or has participated in 2 or more interventional clinical studies in the previous 1 year, or is currently enrolled in any drug or non-drug interventional study.
16. Venous blood concentration of C-reactive protein, measured by high sensitivity assay (hs-CRP) less than 1 mg/L.
17. Has had major surgery, (i.e. requiring general anaesthesia) within 12 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time they are expected to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in total score on the MADRS scale at week 8 | At baseline and at 8 weeks of treatment
  The Montgomery Asberg Depression Rating Scale (MADRS), a researcher-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
  (Visit 4)

SECONDARY OUTCOMES:
Change from baseline in total score on the MADRS scale | At baseline, 2 and 5 weeks of treatment
  The Montgomery Asberg Depression Rating Scale (MADRS), a researcher-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
Change in scores on Perceived Stress Scale | At baseline, 2, 5 and 8 weeks of treatment
  Perceived Stress Scale is a questionnaire measure of recent or current social stress. This scale ranges from 0 to 40; scores ranging from 0-13 would be considered low stress; scores ranging from 14-26 would be considered moderate stress; scores ranging from 27-40 would be considered high perceived stress.
Change in scores on SHAPS | At baseline, 2, 5 and 8 weeks of treatment
  Snaith-Hamilton Pleasure Scale. SHAPS is an instrument developed for the assessment of hedonic capacity and consists of 14-items. Four major domains are covered in the scale, namely interest/pastimes, social interaction, sensory experience, and food/drink. The score range is 0-14. The higher the score the lower the ability to experience pleasure of the patient.
Change in scores on CFQ | At baseline, 2, 5 and 8 weeks of treatment
  Chalder Fatigue Questionnaire (CFQ). The Fatigue Scale, sometimes referred to as the Chalder Fatigue Questionnaire, is a self-administered questionnaire for measuring the extent and severity of fatigue within both clinical and non-clinical, epidemiological populations. The respondent's global score can range from 0 to 33. The global score also spans two dimensions-physical fatigue (measured by items 1-7) and psychological fatigue (measured by items 8-11).
Change in scores on QIDS-SR16 | At baseline, 2, 5 and 8 weeks of treatment
  Quick Inventory of Depressive Symptomatology (QIDS-SR16). The QIDS-SR16 is designed to assess the severity of depressive symptoms and is sensitive to change due to with medications, psychotherapy, or other treatments. Participants will provide responses to each item of this instrument with a 4-point Likert scale, with scores ranging from 0-3 for each item. The total score ranges from 0 to 27. Using a scale of severity of depression of none, mild, moderate, severe, and very severe, corresponding QIDS-SR16 total scores are none 1 to 5, mild 6 to 10, moderate 11 to 15, severe 16 to 20 and very severe 21 to 27.
Change in scores on GAD-7 | At baseline, 2, 5 and 8 weeks of treatment
  Generalized Anxiety Disorder 7 (GAD-7). GAD-7 is a self-reported questionnaire for screening and severity measuring of GAD. GAD-7 has seven items, which measure severity of various signs of GAD according to reported response categories with assigned points. Assessment is indicated by the total score, which made up by adding together the scores for all 7 items. The score ranges from 0 to 21. Using a scale of severity of anxiety of none, mild, moderate and severe, corresponding to GAD-7 total scores are none 0 to 4, mild 5 to 9, moderate 10 to 14 and severe 15 to 21.
Change in score on participant self-reported depression scale | At baseline and at 8 weeks of treatment
  Participants will be asked to self-assess their depression using the Beck Depression Inventory scale (BDI). BDI is a 21-question multiple-choice self-report inventory, widely used for assessment of depression, including in the NIMA BIODEP study, with a score range of 0-63. Each of the 21 items is rated by the participant on a 4 point scale.
Change in scores in the cognitive function test ReVeRe-D | At baseline, 2, 5 and 8 weeks of treatment
  Revere-D is an application developed by Johnson and Johnson, and consists of a battery of eight validated cognitive tasks that assesses cognitive functions, such as memory and learning, that do not involve cognitive processing of emotionally salient stimuli.
Change in scores in Continuous performance test | At baseline, 2, 5 and 8 weeks of treatment
  The continuous performance test is a computerised test of sustained attention which provides a measure of cognitive fatigue.
Change in scores in Emotional Test battery | At baseline and 2 weeks of treatment
  The emotional test battery will consist of 3 validated computerised tasks which are used to assess cognitive functions that involve processing emotionally salient stimuli, such as human faces expressing emotional states.
Change in Brain structure and function | Baseline and at 8 weeks fo treatment
  Brain structure and function will be assessed using fMRI/MRI
Change in heart rate variability | Baseline and at 8 weeks fo treatment
  Heart rate variability will be measured for 15 minutes during rest and whilst completing one of the cognitive tasks.

OTHER OUTCOMES:
Change in Salivary cortisol levels as a measure of biological stress | Samples collected within 7 days prior to Baseline visit and within 7 days prior to visit 4
  Participants will be asked to provide saliva samples before treatment commencement and during the last week of treatment in order for the cortisol levels to be analysed.
Measurement of peripheral blood peripheral cytokine and chemokine levels | Baseline and at 8 weeks fo treatment
  Blood samples will be collected for the analysis of cytokine and chemokine levels with a multiplex immunoassay using the MSD Multi-spot assay system with the Cytokine Panel 1, Proinflammatory panel 1 and Chemokine panel 1 kits providing concentration of all analytes of the panel in pg/ml.
Measurement of peripheral blood immunophenotypes | Baseline and at 8 weeks fo treatment
  The immune cellular content of the blood samples will be analysed with mass cytometry using the commercial kit Maxpar® Direct™ Immune Profiling Assay.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Bullmore, Principal Investigator — Cambridgeshire and Peterborough NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Addenbroooke's Hospital, Cambridge, Cambridgeshire
  - Cardiff University Brain Research Imaging Centre, Cardiff
  - Queen Elizabeth University Hospital, Glasgow
  - The Maurice Wohl Clinical Neuroscience Institute, London
  - Warneford Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
All publications resulting from this study will be made available Open Access. There are plans for anonymised datasets from the trial to become 'open data' and be stored in an online database so that it is publicly available. This page will be updated with information about research outputs as soon as they become available.
Time Frame: After declaration of end of trial to authorities and submission of end of trial report.
Access Criteria: Data will be made available free of charge to anyone interested in the research.